CLINICAL TRIAL: NCT02153983
Title: Pilot Study of the Effects of Colchicine in Non-Diabetic Adults With Metabolic Syndrome
Brief Title: Effects of Colchicine in Non-Diabetic Adults With Metabolic Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jack Yanovski, M.D., Chief, Section on Growth and Obesity, Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 140119; 14-CH-0119 (Other: NIH Clinical Center Protocol Number); ZIAHD000641-23 (NIH)
Record Dates: First submitted 2014-05-31; First posted 2014-06-03 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Obesity; Metabolic Disease
Keywords: Obesity; Colchicine; Inflammation; Metabolic Syndrome; Dyslipidemia
MeSH Terms: conditions — Obesity; Metabolic Diseases; Inflammation; Metabolic Syndrome; Dyslipidemias | interventions — Colchicine; Capsules

STUDY DESIGN:
Intervention Model Description: Note that only 2 of the arms are randomized. Three arms are observational and one is open-label treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In the randomized portion of the trial, all participants, Study Site staff, and pathology and laboratory personnel are blinded to the individual assignment of the order in which colchicine and placebo are administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Obese Adults with Metabolic Syndrome Randomized to Placebo (Experimental): Experimental treatment with placebo capsules identical in appearance to the experimental colchicine preparation
  Interventions: Drug: Placebo capsules given
- Obese Adults with Metabolic Syndrome Randomized to Colchicine (Experimental): Experimental treatment with colchicine capsules identical in appearance to the experimental placebo preparation
  Interventions: Drug: Colchicine 0.6Mg Cap
- Diet-controlled Type 2 Diabetes Adults Assigned to Colchicine (Experimental): Participants with Diet-controlled Type 2 Diabetes who were assigned to Open-label treatment with colchicine. These participants were not randomized and were not part of the randomized controlled trial.
  Interventions: Drug: Colchicine 0.6Mg Tab
- Evaluation Only Non-obese Adults (No Intervention): Participants without obesity seen only for the evaluation component of the study. Such participants are a control group for cross-sectional analyses of baseline data from the experimental cohort.
- Evaluation Only Obese Adults Not Randomized (No Intervention): Participants with obesity seen only for the evaluation component of the study. Such participants are a control group for cross-sectional analyses of baseline data from the experimental cohort. These participants were found not eligible for randomization.
- Evaluation Only Adults with Type 2 Diabetes (No Intervention): Participants with Diet-controlled Type 2 Diabetes seen only for the evaluation component of the study. Such participants are a control group for cross-sectional analyses of baseline data from the experimental cohort.

INTERVENTIONS:
Drug: Colchicine 0.6Mg Cap — Colchicine 0.6 mg given twice daily
  Other Names: RCT Colchicine
  Arms: Obese Adults with Metabolic Syndrome Randomized to Colchicine
Drug: Placebo capsules given — Placebo capsules given twice daily
  Other Names: RCT Placebo
  Arms: Obese Adults with Metabolic Syndrome Randomized to Placebo
Drug: Colchicine 0.6Mg Tab — Open-label colchicine
  Other Names: Open-Label Colchicine 0.6 mg given twice daily
  Arms: Diet-controlled Type 2 Diabetes Adults Assigned to Colchicine

SUMMARY:
Background:

- Being overweight may cause low-level inflammation. This inflammation may cause some of the medical problems of obesity, like high blood sugar (diabetes) and heart disease. This study will test whether a medication called colchicine can improve metabolism in adults who are overweight but have not yet developed diabetes.

Objectives:

- To learn whether colchicine improves sugar regulation and metabolism.

Eligibility:

- Healthy overweight adults18 to 100 years old.

Design:

* Participants must fast before each visit, including the screening visit.
* Participants will be screened with blood tests,urine tests, medical history, and physical exam. They will have to drink sugar water, and have blood drawn to find out if they are healthy.
* For visit 1, participants will have a medical history and physical exam and answer questions. They will have blood taken with an intravenous (IV) line, give urine sample, and give 2 stool samples..
* Also, subjects will get sugar water through one IV. Blood will be drawn from the other. This measures sugar and insulin levels. During this, participants will lie in a bed and can watch TV.
* Participants will have a full-body X-ray, lying on a table while a camera passes over them. They will also have an abdominal CT scan, lying on a table that moves through a ring that takes pictures.
* Participants will have a small fat tissue sample taken from their abdomen. It is like getting a mini-liposuction.
* Participants will be given the study drug or placebo. They will take it twice daily for 3 months.
* For visit 2, participants will have blood tests, urine tests, medical history, and physical exam.
* For visit 3, participants will repeat the tests in visit 1.

DETAILED DESCRIPTION:
Obesity affects one-third of the adult U.S. population and is a major risk factor for the development of type 2 diabetes and cardiovascular disease. Mouse models and human data suggest that obesity-induced chronic inflammation is one mechanism promoting obesity-associated comorbid conditions. In obesity, innate immunity is activated by circulating molecules such as fatty acids and cholesterol crystals bind to nucleotide-binding oligomerization (NOD)-like receptor family, pyrin domain containing 3 (NLRP3) receptors in adipocyte tissue macrophages (ATMs). This binding stimulates NLRP3 oligomerization, inflammasome formation, and proinflammatory cytokine activation. The resultant inflammatory cascade leads to insulin resistance and decreased pancreatic beta-cell reserve. It has been proposed that the suppression of this chronic low-level inflammatory state may impede the onset of diabetes and cardiovascular disease.

Recent studies have shown colchicine, a potent microtubule inhibitor commonly used for the treatment of gout and some rare inflammatory conditions, disrupts intracellular localization of NLRP3, thereby blocking inflammasome assembly. As there are limited medical therapies proven effective to improve obesity-related metabolic dysregulation, we propose to determine the efficacy of colchicine 0.6 mg twice daily in non-diabetic obese adults with metabolic syndrome. We will conduct a randomized, double-blinded, placebo-controlled pilot trial of colchicine in forty subjects. We will study changes in insulin resistance, beta-cell reserve, and systemic inflammation. Using adipose tissue obtained from biopsies, we will also study colchicine s local effects on inflammation and insulin resistance. Should results prove promising, this pilot study will allow determination of the sample size needed for an adequately powered study of the effects of colchicine in obese adults with metabolic syndrome.

Seven patients with diet-controlled type 2 diabetes will be given open-label colchicine and followed as described above. We also plan to perform baseline evaluations on 40 subjects who are not eligible for the treatment protocol. This group will consist of non-obese adults, obese adults who are not insulin-resistant, and adults with diet-controlled type 2 diabetes.

ELIGIBILITY:
* INCLUSION CRITERIA FOR SUBJECTS RANDOMIZED TO COLCHICINE or PLACEBO::

Subjects will qualify for randomization to colchicine or placebo if they meet the following criteria:

* Good general health. In general subjects should take no medications. However, individuals taking medications for obesity-related co-morbid conditions, who have not had changes in dosage for more than 3 months, may be included, at the discretion of the principal investigator.
* Obesity, defined as a body mass index (BMI) greater than or equal to 30 kg/m^2, but weight less than 450 lbs in order for subjects to undergo Dual-Energy X-ray Absorptiometry (DXA) scanning.
* Age 18 to 100 years.
* Metabolic Syndrome defined as any 3 of the following 5:

  * FPG greater than or equal to 100 mg/dl, or Impaired Glucose Tolerance (Glucose greater than or equal to 140 mg/dl at 2 hours of OGTT)
  * Triglycerides greater than or equal to 150 mg/dl, or on treatment
  * Waist Circumference: Men greater than or equal to 40 in (greater than or equal to 102 cm); Women greater than or equal to 35 in (greater than or equal to 88 cm)
  * Reduced HDL-C: Men < 40 mg/dl; Women < 50 mg/dl, or on treatment
  * Hypertension: greater than or equal to 130 mmHg systolic, or greater than or equal to 85 mmHg diastolic, or on treatment
* HOMA-IR greater than or equal to 2.6. Our goal is to enroll participants who have pre-existing insulin resistance.
* high sensitivity C-reactive protein (hs-CRP) greater than or equal to 2.0 mg/L. We aim to recruit participants with increased baseline level of inflammation. Individuals with hsCRP above 2.0 mg/L have been shown to have an increased risk for cardiovascular events.

EXCLUSION CRITERIA FOR SUBJECTS RANDOMIZED TO COLCHICINE OR PLACEBO:

* Type 2 diabetes mellitus, as determined by either having:

  * Clear clinical diagnosis of diabetes, such as a patient in a hyperglycemic crisis or classic symptoms of hyperglycemia and a random plasma glucose greater than or equal to 200 mg/dL
  * Two of the following three:

    * Fasting plasma glucose greater than or equal to 126 mg/dL
    * Hemoglobin A1c greater than or equal to 6.5%
    * An oral glucose tolerance test glucose concentration of greater than or equal to 200 mg/dL at 2 hours.
  * One of the above three criteria (bi.-biii.) meeting the T2DM cutoff on two different days. If only one of the above three criteria (bi.-biii.) meet the T2DM threshold during the Screening Visit, that test will be repeated on another day to determine if the subject has T2DM or not. As per ADA guidelines, The diagnosis [of T2DM] is made on the basis of the confirmed test.Moreover, because HbA1c has been shown to be higher in African Americans (AA) as compared to other races for the same glycemia, non-diabetic AA may be unfairly excluded by their HbA1c alone. Therefore, for AA subjects, if their 2 hour OGTT and fasting glucoses are in the non-diabetic range, and the HbA1c is < 7.0%, we will consider them non-diabetic.
* Presence of a significant active or chronic illness likely to limit life span and/or increase risk of intervention, including renal (GFR less than or equal to 60 ml/min/1.73m2), cardiovascular, hepatic (other than obesity-related steatosis), gastrointestinal, immunologic, endocrinologic (e.g. Cushing syndrome), pulmonary (other than either asthma not requiring continuous medication or sleep apnea-related disorders), or other disorders at the discretion of the investigators.
* Recent use of colchicine or anorexiant medications in the last 3 months.
* Known allergy to colchicine.
* Previous history of agranulocytosis, gout, or significant myositis.
* Females who are pregnant, planning to become pregnant, currently nursing an infant, or have irregular menses, defined as cycles less than 21 days or greater than 45 days.
* Individuals who have current substance abuse or a psychiatric disorder or any other condition that in the opinion of the investigators would impede competence, compliance, or participation in the study.
* Subjects who regularly use prescription medications unrelated to the complications of obesity, especially those known to affect enzymes involved in colchicine metabolism, such as CYP3A4 or P-glycoprotein (P-gp) . Oral contraceptive use will be permitted, provided the contraceptive has been used for at least two months before starting study medication. The use of over-the-counter and prescription medications will be reviewed on a case-by-case basis; depending on the medication, subjects who have continued to take prescription medication or have stopped taking an exclusionary medication for at least 3 months prior to study entry may be eligible .
* Participation in a formal weight loss program (e.g. Weight Watchers) or recent weight change of more than 3% of body weight in the past two months.
* Use of anti-inflammatory medications (e.g. prednisone, NSAIDs) chronically or in the last 7 days prior to fat biopsy.
* History of keloid formation.
* Current users of tobacco or nicotine products (e.g. nicotine patch, e-cigarettes).

INCLUSION CRITERIA FOR SUBJECTS WHO ARE EVALUATED BUT NOT ELIGIBLE FOR RANDOMIZATION:

Subjects will qualify for the Evaluation-only arm if they meet the following criteria:

* Good general health. In general subjects should take no medications. The use of over-the-counter and prescription medications will be reviewed on a case-by-case basis; depending on the medication, subjects who have continued to take prescription medication or have stopped taking an exclusionary medication for at least 3 months prior to study entry may be eligible.
* Weight less than 450 lbs in order for subjects to undergo Dual-Energy X-ray Absorptiometry (DXA) scanning.
* Age 18 years to 100 years.

EXCLUSION CRITERIA FOR SUBJECTS WHO ARE EVALUATED BUT NOT ELIGIBLE FOR RANDOMIZATION:<TAB>

* Type 2 diabetes mellitus that is not well controlled with diet alone: subjects taking an antidiabetic medication (e.g. metformin, insulin, sulfonylureas, etc.) or having a Hemoglobin A1c > 9.0%
* Presence of a significant active or chronic illness likely to limit life span and/or increase risk of intervention, including renal (GFR less than or equal to 60 ml/min/1.73m2), cardiovascular, hepatic (other than obesity-related steatosis), gastrointestinal, immunologic, endocrinologic (e.g. Cushing syndrome), pulmonary (other than either asthma not requiring continuous medication or sleep apnea-related disorders), or other disorders at the discretion of the investigators.
* Recent use of colchicine or anorexiant medications in the last 3 months.
* Females who are pregnant, planning to become pregnant, or are currently nursing an infant.
* Individuals who have current substance abuse or a psychiatric disorder or any other condition that in the opinion of the investigators would impede competence, compliance, or participation in the study.
* Participation in a formal weight loss program (e.g. Weight Watchers) or recent weight change of more than 3% of body weight in the past two months.
* Use of anti-inflammatory medications (e.g. prednisone, NSAIDs) chronically or in the last 7 days prior to fat biopsy.
* History of keloid formation.
* Current users of tobacco or nicotine products (e.g. nicotine patch, e-cigarettes).

INCLUSION CRITERIA FOR SUBJECTS WITH DIET-CONTROLLED T2DM

Subjects will qualify for the Open Label arm if they meet the following criteria:

* A diagnosis of T2DM.

  * Not on any diabetic/hypoglycemic agents
  * Not having an alternate cause of hyperglycemia (e.g. T1DM, glucocorticoidinduced, lipodystrophy, acromegaly, etc.)
* Hemoglobin A1c less than or equal to 9.0%
* Good general health. In general subjects should take no medications. The use of over-the-counter and prescription medications will be reviewed on a case-by-case basis; depending on the medication, subjects who have continued to take prescription medication or have stopped taking an exclusionary medication for at least 3 months prior to study entry may be eligible
* Age greater than or equal to 18 to 100 years.
* Obesity, defined as a body mass index (BMI) greater than or equal to 30 kg/m2, but weight less than 450 lbs in order for subjects to undergo Dual-Energy X-ray Absorptiometry (DXA) scanning.
* Metabolic Syndrome

(Any 3 of the following 5):

* FPG greater than or equal to100 mg/dl or Impaired Glucose Tolerance (Glucose greater than or equal to 140 mg/dl at 2 hours of OGTT)
* Triglycerides greater than or equal to 150 mg/dl, or on treatment
* Waist Circumference: Men greater than or equal to 40 in (greater than or equal to 102 cm); Women greater than or equal to 35 in (greater than or equal to 88 cm)
* Reduced HDL-C: Men < 40 mg/dl; Women < 50 mg/dl, or on treatment
* Hypertension: greater than or equal to 130 mmHg systolic, or greater than or equal to 85 mmHg diastolic, or on treatment

  * HOMA-IR greater than or equal to 2.6. Our goal is to enroll participants who have pre-existing insulinresistance.
  * hsCRP greater than or equal to 2.0 mg/L. We aim to recruit participants with increased baseline level of inflammation. Individuals with hsCRP above 2.0 mg/L have been shown to have an increased risk for cardiovascular events.

EXCLUSION CRITERIA FOR SUBJECTS WITH DIET-CONTROLLED T2DM

* T2DM that is not well controlled with diet alone: subjects will not be eligible if they take an anti-diabetic medication (e.g. metformin, insulin, sulfonylurea, etc.), or have HbA1c >9%.
* Presence of a significant active or chronic illness likely to limit life span and/or increase risk of intervention, including renal (GFR less than or equal to 30 ml/min/1.73m2), cardiovascular, hepatic (other than obesity-related steatosis), gastrointestinal, immunologic, endocrinologic (e.g. Cushing syndrome), pulmonary (other than either asthma not requiring continuous medication or sleep apnea-related disorders), or other disorders at the discretion of the investigators.
* Recent use of colchicine or anorexiant medications in the last 3 months.
* Known allergy to colchicine.
* Previous history of agranulocytosis, gout, or significant myositis.
* Females who are pregnant, planning to become pregnant, currently nursing an infant, or have irregular menses, defined as cycles less than 21 days or greater than 45 days.
* Individuals who have current substance abuse or a psychiatric disorder or any other condition that in the opinion of the investigators would impede competence, compliance, or participation in the study.
* Subjects who regularly use prescription medications unrelated to the complications of obesity, especially those known to affect enzymes involved in colchicine metabolism, such as CYP3A4 or P-glycoprotein (P-gp). Oral contraceptive use will be permitted, provided the contraceptive has been used for at least two months before starting study medication. The use of over-the-counter and prescription medications will be reviewed on a case-by-case basis; depending on the medication, subjects who have continued to take prescription medication or have stopped taking an exclusionary medication for at least 3 months prior to study entry may be eligible.
* Participation in a formal weight loss program (e.g. Weight Watchers) or recent weight change of more than 3% of body weight in the past two months.
* Use of anti-inflammatory medications (e.g. prednisone, NSAIDs) chronically or in the last 7 days prior to fat biopsy.
* History of keloid formation.
* Current users of tobacco or nicotine products (e.g. nicotine patch, e-cigarettes).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-05-31; Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Yanovski, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual-level data for the primary and secondary outcomes will be made available upon request. PII will be removed.
Supporting Information: Study Protocol, ICF
Time Frame: in July 2021, and then indefinitely
Access Criteria: Approval of the PI
URL: https://dash.nichd.nih.gov/

REFERENCES:
- [Background] Wen H, Gris D, Lei Y, Jha S, Zhang L, Huang MT, Brickey WJ, Ting JP. Fatty acid-induced NLRP3-ASC inflammasome activation interferes with insulin signaling. Nat Immunol. 2011 May;12(5):408-15. doi: 10.1038/ni.2022. Epub 2011 Apr 10. PMID 21478880
- [Background] Vandanmagsar B, Youm YH, Ravussin A, Galgani JE, Stadler K, Mynatt RL, Ravussin E, Stephens JM, Dixit VD. The NLRP3 inflammasome instigates obesity-induced inflammation and insulin resistance. Nat Med. 2011 Feb;17(2):179-88. doi: 10.1038/nm.2279. Epub 2011 Jan 9. PMID 21217695
- [Background] Demidowich AP, Davis AI, Dedhia N, Yanovski JA. Colchicine to decrease NLRP3-activated inflammation and improve obesity-related metabolic dysregulation. Med Hypotheses. 2016 Jul;92:67-73. doi: 10.1016/j.mehy.2016.04.039. Epub 2016 Apr 25. PMID 27241260
- [Result] Demidowich AP, Levine JA, Onyekaba GI, Khan SM, Chen KY, Brady SM, Broadney MM, Yanovski JA. Effects of colchicine in adults with metabolic syndrome: A pilot randomized controlled trial. Diabetes Obes Metab. 2019 Jul;21(7):1642-1651. doi: 10.1111/dom.13702. Epub 2019 Apr 2. PMID 30869182
- [Derived] Levine JA, Han JM, Wolska A, Wilson SR, Patel TP, Remaley AT, Periwal V, Yanovski JA, Demidowich AP. Associations of GlycA and high-sensitivity C-reactive protein with measures of lipolysis in adults with obesity. J Clin Lipidol. 2020 Sep-Oct;14(5):667-674. doi: 10.1016/j.jacl.2020.07.012. Epub 2020 Aug 4. PMID 32863171
- [Derived] Demidowich AP, Wolska A, Wilson SR, Levine JA, Sorokin AV, Brady SM, Remaley AT, Yanovski JA. Colchicine's effects on lipoprotein particle concentrations in adults with metabolic syndrome: A secondary analysis of a randomized controlled trial. J Clin Lipidol. 2019 Nov-Dec;13(6):1016-1022.e2. doi: 10.1016/j.jacl.2019.10.011. Epub 2019 Oct 22. PMID 31740368
- [Derived] Demidowich AP, Parikh VJ, Dedhia N, Branham RE, Madi SA, Marwitz SE, Roberson RB, Uhlman AJ, Levi NJ, Mi SJ, Jun JY, Broadney MM, Brady SM, Yanovski JA. Associations of the melanocortin 3 receptor C17A + G241A haplotype with body composition and inflammation in African-American adults. Ann Hum Genet. 2019 Sep;83(5):355-360. doi: 10.1111/ahg.12315. Epub 2019 Apr 2. PMID 30937899
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-CH-0119.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 213 adults were screened in the clinic and signed consent forms, of whom 77 were found eligible and studied with protocols.
Groups:
- Obese Adults With Metabolic Syndrome Randomized to Placebo: Experimental treatment with placebo capsules identical in appearance to the experimental colchicine preparation given twice daily
- Obese Adults With Metabolic Syndrome Randomized to Colchicine: Experimental treatment with colchicine capsules identical in appearance to the experimental placebo preparation given twice daily
- Open Label Patients With Type 2 Diabetes: Patients with diet-controlled type 2 dabetes, given open-label colchicine tablets 0.6 mg twice-daily
- Evaluation Only Non-obese Adults: Adults without obesity, seen only for an evaluation visit, not given any medication and not followed longitudinally.
- Evaluation Only Obese Adults: Adults with obesity, seen only for an evaluation visit, not given any medication and not followed longitudinally.
- Evaluation Only Adults With Type 2 Diabetes: Adults with Diet-controlled Type 2 Diabetes, seen only for an evaluation visit, not given any medication and not followed longitudinally.
Period: Overall Study
Arm/Group | Obese Adults With Metabolic Syndrome Randomized to Placebo | Obese Adults With Metabolic Syndrome Randomized to Colchicine | Open Label Patients With Type 2 Diabetes | Evaluation Only Non-obese Adults | Evaluation Only Obese Adults | Evaluation Only Adults With Type 2 Diabetes
Started | 19 | 21 | 4 | 13 | 19 | 1
Completed | 19 | 18 | 2 | 13 | 19 | 1
Not Completed | 0 | 3 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants are adults with high C-reactive protein, obesity, and metabolic syndrome. Open-label patients have Type 2 diabetes. Evaluation Only participants did not have to have obesity, diabetes, metabolic syndrome, or high C-reactive protein.
Groups:
- Open Label Patients With Type 2 Diabetes: Adults with diet-controlled type 2 diabetes, treated with open-label Colchicine 0.6Mg Tab
- Evaluation Only Adults With Diet-controlled Type 2 Diabetes: Adults with Diet-controlled Type 2 Diabetes, seen only for an evaluation visit, not given any medication and not followed longitudinally.
- Total: Total of all reporting groups
Arm/Group | Obese Adults With Metabolic Syndrome Randomized to Placebo | Obese Adults With Metabolic Syndrome Randomized to Colchicine | Open Label Patients With Type 2 Diabetes | Evaluation Only Non-obese Adults | Evaluation Only Obese Adults | Evaluation Only Adults With Diet-controlled Type 2 Diabetes | Total
Number analyzed (Participants) | 19 | 21 | 4 | 13 | 19 | 1 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (10.0) | 47.3 (13.4) | 42.8 (13.4) | 37.2 (13.5) | 46.4 (11.9) | 47.9 | 44.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 4 | 8 | 15 | 0 | 58
  Male | 4 | 5 | 0 | 5 | 4 | 1 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 3 | 1 | 3 | 0 | 19
  Not Hispanic or Latino | 12 | 15 | 1 | 11 | 16 | 1 | 56
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 1 | 3 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 6 | 1 | 6 | 5 | 1 | 24
  White | 7 | 9 | 0 | 4 | 8 | 0 | 28
  More than one race | 2 | 2 | 0 | 1 | 0 | 0 | 5
  Unknown or Not Reported | 4 | 3 | 3 | 1 | 3 | 0 | 14
High-Sensitivity C-Reactive Protein [Mean (Standard Deviation); unit: mg/L] | 6.7 (4.2) | 8.1 (7.4) | 9.63 (6.17) | 0.77 (0.80) | 3.08 (2.67) | 1.4 | 5.41 (5.49)

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Sensitivity From FSIVGTT
Description: Change (3 month minus minus baseline) in insulin sensitivity value, calculated from frequently-sampled intravenous glucose tolerance tests by Bergman's Minimal Model using intent-to-treat. Higher values represent a better outcome. There are no data from the evaluation-only participants, since they were not followed longitudinally.
Time Frame: Baseline to 3 months
Population: Randomized trial has 2 groups, open label only one group
Measure: Mean (95% Confidence Interval); unit: 10^-5*min^-1*mU^-1*mL
Groups:
- Obese Adults With Metabolic Syndrome Randomized to Placebo: Experimental treatment with placebo capsules identical in appearance to the experimental colchicine preparation, given twice daily
- Open Label Patients With Type 2 Diabetes: Patients With Type 2 Diabetes given open-label treatment with colchicine 0.6 Mg Tab
Arm/Group | Obese Adults With Metabolic Syndrome Randomized to Placebo | Obese Adults With Metabolic Syndrome Randomized to Colchicine | Open Label Patients With Type 2 Diabetes
Number analyzed (Participants) | 19 | 21 | 4
10^-5*min^-1*mU^-1*mL | 0.20 [-0.12 to 1.58] | 0.41 [-0.90 to 1.72] | -0.45 [-1.58 to 0.61]

2. Secondary Outcome: Change in HOMA-IR Index
Description: Change (3 month minus minus baseline) in calculated homeostasis model of insulin sensitivity, calculated from derived from fasting glucose and insulin values = fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5) using intent-to-treat. Higher values represent a worse outcome. There are no data from the evaluation-only participants, since they were not followed longitudinally.
Time Frame: Baseline to 3 months
Population: RCT has colchicine and placebo groups, open label is colchicine only.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Open Label Patients With Type 2 Diabetes: Patients With Type 2 Diabetes given open-label colchicine tablets twice daily.
Arm/Group | Obese Adults With Metabolic Syndrome Randomized to Placebo | Obese Adults With Metabolic Syndrome Randomized to Colchicine | Open Label Patients With Type 2 Diabetes
Number analyzed (Participants) | 19 | 21 | 4
units on a scale | 1.1 [-0.1 to 7.6] | -0.3 [-1.1 to 1.1] | 8.4 [0.05 to 16.8]

3. Secondary Outcome: Changes in C-reactive Protein
Description: Change (3 month minus minus baseline) in High-Sensitivity C-reactive protein concentrations using intent-to-treat. Higher values represent a worse outcome. There are no data from the evaluation-only participants, since they were not followed longitudinally.
Time Frame: Baseline to 3 months
Population: Patients randomized to colchicine or placebo for randomized controlled trial, but only open-label colchicine for patients with type 2 diabetes
Measure: Mean (95% Confidence Interval); unit: mg/L
Groups:
- Open Label Patients With Type 2 Diabetes: Patients with type 2 diabetes given open-label colchicine tablets
Arm/Group | Obese Adults With Metabolic Syndrome Randomized to Placebo | Obese Adults With Metabolic Syndrome Randomized to Colchicine | Open Label Patients With Type 2 Diabetes
Number analyzed (Participants) | 19 | 21 | 4
mg/L | 0.5 [-0.9 to 1.8] | -2.8 [-4.1 to -1.5] | -3.7 [-10.4 to 3.0]

ADVERSE EVENTS:
Time Frame: 3 months of treatment
Groups:
- Open Label Patients With Type 2 Diabetes: Open-label treatment with colchicine
  Colchicine 0.6Mg Tab: Open-label colchicine
- Evaluation Only Non-obese Adults: No treatment non-obese adults seen only for evaluation
- Evaluation Only Obese Adults: No treatment obese adults seen only for evaluation
- Evaluation Only Adults With Diet-controlled Type 2 Diabetes: No treatment adults with Type 2 Diabetes seen only for evaluation
Arm/Group | Obese Adults With Metabolic Syndrome Randomized to Placebo | Obese Adults With Metabolic Syndrome Randomized to Colchicine | Open Label Patients With Type 2 Diabetes | Evaluation Only Non-obese Adults | Evaluation Only Obese Adults | Evaluation Only Adults With Diet-controlled Type 2 Diabetes
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21 | 0/4 | 0/13 | 0/19 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21 | 0/4 | 0/13 | 0/19 | 0/1
Other Adverse Events (participants affected / at risk) | 16/19 | 15/21 | 2/4 | 0/13 | 0/19 | 0/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obese Adults With Metabolic Syndrome Randomized to Placebo (N=19) | Obese Adults With Metabolic Syndrome Randomized to Colchicine (N=21) | Open Label Patients With Type 2 Diabetes (N=4) | Evaluation Only Non-obese Adults (N=13) | Evaluation Only Obese Adults (N=19) | Evaluation Only Adults With Diet-controlled Type 2 Diabetes (N=1)
Gastrointestinal (Gastrointestinal disorders) | 14 (14) | 13 (13) | 1 (4) | 0 (0) | 0 (0) | 0 (0) — Nausea, vomiting, or diarrhea
Upper Respiratory Tract (Infections and infestations) | 11 (11) | 6 (6) | 1 (4) | 0 (0) | 0 (0) | 0 (0) — Viral syndrome, Upper Respiratory Illness
Fatigue (General disorders) | 5 (5) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated Creatine Kinase (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated Alanine Aminotransferase (Hepatobiliary disorders) | 2 (2) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated Aspartate Aminotransferase (Hepatobiliary disorders) | 4 (4) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Pilot trial to determine power calculations, so no definitive conclusions should be reached from this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/83/NCT02153983/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/83/NCT02153983/ICF_001.pdf